CLINICAL TRIAL: NCT04232566
Title: Investigating the Link Between Type 2 Immunity and NAFLD in Human Obesity- AIM 1
Brief Title: Investigating the Link Between Type 2 Immunity and NAFLD in Human Obesity
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elena Anna (Eleanna) De Filippis, M.D., Ph.D., Principal Investigator, Mayo Clinic
Other Study IDs: 18-004615
Record Dates: First submitted 2019-01-02; First posted 2020-01-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity, Morbid; NASH - Nonalcoholic Steatohepatitis; Chronic Inflammation
Keywords: obesity; nash; adipose tissue inflammation; insulin resistance
MeSH Terms: conditions — Obesity, Morbid; Non-alcoholic Fatty Liver Disease; Obesity; Insulin Resistance | interventions — Bariatric Surgery; Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Weight loss surgery: Gastric bypass surgery will be followed by weight loss as standard of care. Liver fibrosis by elastography will be determined before surgery.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Evaluate liver fibrosis by elastography before gastric bypass surgery.
  Other Names: Roux en Y gastric bypass, sleeve gastrectomy

SUMMARY:
This study is being done to better understand the relationship between inflammation in adipose tissue (AT), abnormal deposition of fat around the liver and how this affects its appearance and function and ultimately insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing gastric bypass surgery
* Confirmed AUROC F=0 or F>2 liver fibrosis
* Age 30-70 years
* BMI greater than 40 kg/m2
* Negative pregnancy test (female only)
* Lab Values: Normal TSH

Exclusion Criteria:

* Autoimmune diseases
* Hepatitis B or C positive
* Heavy alcohol use
* Active smoking history
* Active cancer history
* History of asthma
* History of COPD
* Taking Plavix or Coumadin
* Blood donation within past 2 months
* Glucocorticoid Therapy
* Taking antihistamine on regular basis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fourteen subjects with F=0 (no fibrosis) and forty-six patients undergoing gastric bypass Surgery with confirmed Area under the Receiver Operating Characteristic Curve (AUROC) F>2 (moderate fibrosis), age 30-70yrs, both genders, BMI greater than 40 kg/m2 will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Liver fibrosis | Baseline
  evaluate the liver fibrosis by elastography before surgical intervention
Adipose tissue inflammation | Baseline
  Evaluate markers of adipose tissue inflammation by mRNA levels

CONTACTS AND LOCATIONS:
Overall Officials: Elena Anna O De Filippis, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No